CLINICAL TRIAL: NCT05779670
Title: Treatment Adherence to a Personalized Home Exercise Program in Patients With Bone Cancer Undergoing Lower Extremity Resection and Reconstruction
Brief Title: Adherence to a Personalized Home Exercise Program in Patients With Bone Tumor Undergoing Lower Extremity Salvage Surgery
Acronym: ADER
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 5001
Record Dates: First submitted 2023-03-06; First posted 2023-03-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Osteosarcoma; Ewing Sarcoma; Chondrosarcoma; Bone Tumor
Keywords: rehabilitation; home based exercise; bone tumor
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing; Chondrosarcoma; Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to describe adherence to a personalised home exercise program in patients undergoing resection and reconstruction of lower limb for bone tumor and neoadjuvant chemotherapy treatment in the first six months after surgery intervention and investigate possible prognostic factors.

DETAILED DESCRIPTION:
In cancer patients undergoing adjuvant therapies, rehabilitation plays an important role in reducing the side effects of chemotherapy treatment by promoting cardiorespiratory function, reducing fatigue and improving quality of life. Physiotherapy treatment, generally, includes physical training programs administered in many ways, not yet well standardized. With the aim of seeking an empowerment of the patient and his active participation, more and more exercise programs are used that the patient is able to manage independently. Adherence to and compliance with such exercise programs is extremely variable in literature and can range from 52% to 89%. A high level of adhesion is a well-known challenge and a fundamental prerequisite for achieving the benefits of physical activity. Home exercise programs to be performed in complete autonomy have been proposed in patients with different types of cancer, while for patients with bone tumor, to date there are no experiences. In this group of patients the role of physiotherapy is significant not only to counteract the adverse effects of chemotherapy treatment but also to promote the recovery of patients following the important resection and reconstruction interventions. In this type of patient, a high adherence to the physiotherapy treatment started already during the periods of hospitalization for the administration of antiblastic treatment.

Data will be collected from all patients treated consecutively over two years according to the defined inclusion criteria. Given the rarity of oncologic pathology of the musculoskeletal system and the limited number of patients of 27 found to meet the inclusion criteria in the year 2021, it is assumed that data will be collected from a sample of 50 patients.

The variables collected will be: age, sex, BMI, smoking, physical activity level, diagnosis, metastasis at diagnosis, type of surgery, chemotherapy treatment.

Data will be described by mean and standard deviation or median and interquartile range values according to the nature of the data and frequency and percentage for dichotomous variables

The objective of this study is to describe adherence to a personalised home exercise program in patients undergoing resection and reconstruction of lower limb for bone tumor and neoadjuvant chemotherapy treatment in the first six months after surgery intervention and investigate possible prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 12 years with bone tumor undergoing surgery (resection and reconstruction of the lower limb) and in adjuvant treatment
* patients under physiotherapy treatment

Exclusion Criteria:

* patients with difficulties in understanding the Italian language
* patients not using digital services

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Will be recruited consecutively all patients with bone cancer undergoing resection and reconstruction of the lower limb at the "Orthopedic and Traumatological Clinic III to prevalent oncological address" of the Rizzoli Orthopaedic Institute in the period from 01/2023 to 12/2024 and subsequently to the "SC Osteoncologia, sarcomas of bone and soft tissues, and innovative therapies of the same hospital for the continuation of treatment" in the next six months after surgery.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
adherence to the rehabilitation program | everyday from baseline at 6 months
  every day the patient will record the exercise execution/not-execution

SECONDARY OUTCOMES:
TESS | at 3 months and at 6 months
  The TESS is a self-administered questionnaire evaluating possible limitations in physical activity. A total of 30 questions are included in the TESS, and the degree of disability is rated from 0 (complete disability) to 5 (no functional impairment) in each item. Similar to MSTS for lower extremity, the final TESS score is converted to a score ranging from 0 to 100 points. If a question in TESS score does not apply to the patient, the last can respond "not applicable."
TUG | at 3 months and at 6 months
  Timed up and go is a simple test to measure a person's mobility level and requires static and dynamic balancing skills. It consists of measuring how many seconds it takes the patient to get up from the chair, walk a distance of 3 meters, turn around, return to the chair and sit down again.
patient satisfaction | at 3 months and at 6 months
  will be investigated with a questionnaire consisting of a likert scale of 4 questions with score from 0 (not at all satisfied) to 5 (completely satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: alida abbruzzese, Principal Investigator — ufficio ricerca professioni sanitarie
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Cramp F, Byron-Daniel J. Exercise for the management of cancer-related fatigue in adults. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD006145. doi: 10.1002/14651858.CD006145.pub3. PMID 23152233
- [Background] van Weert E, Hoekstra-Weebers JE, May AM, Korstjens I, Ros WJ, van der Schans CP. The development of an evidence-based physical self-management rehabilitation programme for cancer survivors. Patient Educ Couns. 2008 May;71(2):169-90. doi: 10.1016/j.pec.2007.11.027. Epub 2008 Feb 5. PMID 18255249
- [Background] Mishra SI, Scherer RW, Snyder C, Geigle PM, Berlanstein DR, Topaloglu O. Exercise interventions on health-related quality of life for people with cancer during active treatment. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD008465. doi: 10.1002/14651858.CD008465.pub2. PMID 22895974
- [Background] Jones LW, Liang Y, Pituskin EN, Battaglini CL, Scott JM, Hornsby WE, Haykowsky M. Effect of exercise training on peak oxygen consumption in patients with cancer: a meta-analysis. Oncologist. 2011;16(1):112-20. doi: 10.1634/theoncologist.2010-0197. Epub 2011 Jan 6. PMID 21212429
- [Background] Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. JAMA. 2002 Nov 20;288(19):2469-75. doi: 10.1001/jama.288.19.2469. PMID 12435261
- [Background] Mock V, Dow KH, Meares CJ, Grimm PM, Dienemann JA, Haisfield-Wolfe ME, Quitasol W, Mitchell S, Chakravarthy A, Gage I. Effects of exercise on fatigue, physical functioning, and emotional distress during radiation therapy for breast cancer. Oncol Nurs Forum. 1997 Jul;24(6):991-1000. PMID 9243585
- [Background] Schwartz AL. Daily fatigue patterns and effect of exercise in women with breast cancer. Cancer Pract. 2000 Jan-Feb;8(1):16-24. doi: 10.1046/j.1523-5394.2000.81003.x. PMID 10732535
- [Background] Schwartz AL. Exercise and weight gain in breast cancer patients receiving chemotherapy. Cancer Pract. 2000 Sep-Oct;8(5):231-7. doi: 10.1046/j.1523-5394.2000.85007.x. PMID 11898235
- [Background] Segar ML, Katch VL, Roth RS, Garcia AW, Portner TI, Glickman SG, Haslanger S, Wilkins EG. The effect of aerobic exercise on self-esteem and depressive and anxiety symptoms among breast cancer survivors. Oncol Nurs Forum. 1998 Jan-Feb;25(1):107-13. PMID 9460778
- [Background] Pickett M, Mock V, Ropka ME, Cameron L, Coleman M, Podewils L. Adherence to moderate-intensity exercise during breast cancer therapy. Cancer Pract. 2002 Nov-Dec;10(6):284-92. doi: 10.1046/j.1523-5394.2002.106006.x. PMID 12406050
- [Background] Markes M, Brockow T, Resch KL. Exercise for women receiving adjuvant therapy for breast cancer. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD005001. doi: 10.1002/14651858.CD005001.pub2. PMID 17054230
- [Background] Kampshoff CS, Jansen F, van Mechelen W, May AM, Brug J, Chinapaw MJ, Buffart LM. Determinants of exercise adherence and maintenance among cancer survivors: a systematic review. Int J Behav Nutr Phys Act. 2014 Jul 2;11:80. doi: 10.1186/1479-5868-11-80. PMID 24989069
- [Background] American College of Sports Medicine Position Stand. The recommended quantity and quality of exercise for developing and maintaining cardiorespiratory and muscular fitness, and flexibility in healthy adults. Med Sci Sports Exerc. 1998 Jun;30(6):975-91. doi: 10.1097/00005768-199806000-00032. PMID 9624661
- [Background] Lund LW, Ammitzboll G, Hansen DG, Andersen EAW, Dalton SO. Adherence to a long-term progressive resistance training program, combining supervised and home-based exercise for breast cancer patients during adjuvant treatment. Acta Oncol. 2019 May;58(5):650-657. doi: 10.1080/0284186X.2018.1560497. Epub 2019 Jan 30. PMID 30698050
- [Background] Kim JY, Lee MK, Lee DH, Kang DW, Min JH, Lee JW, Chu SH, Cho MS, Kim NK, Jeon JY. Effects of a 12-week home-based exercise program on quality of life, psychological health, and the level of physical activity in colorectal cancer survivors: a randomized controlled trial. Support Care Cancer. 2019 Aug;27(8):2933-2940. doi: 10.1007/s00520-018-4588-0. Epub 2018 Dec 18. PMID 30564936
- [Background] Nyrop KA, Deal AM, Choi SK, Wagoner CW, Lee JT, Wood WA, Anders C, Carey LA, Dees EC, Jolly TA, Reeder-Hayes KE, Muss HB. Measuring and understanding adherence in a home-based exercise intervention during chemotherapy for early breast cancer. Breast Cancer Res Treat. 2018 Feb;168(1):43-55. doi: 10.1007/s10549-017-4565-1. Epub 2017 Nov 9. PMID 29124455
- [Background] Wang YQ, Liu X, Yin YY, Ma RC, Yang Z, Cao HP, Xie J. Effects of Home-Based Exercise Training for Patients With Lung Cancer. Oncol Nurs Forum. 2019 Jul 1;46(4):E119-E134. doi: 10.1188/19.ONF.E119-E134. PMID 31225844
- [Background] van Waart H, Buffart LM, Stuiver MM, van Harten WH, Sonke GS, Aaronson NK. Adherence to and satisfaction with low-intensity physical activity and supervised moderate-high intensity exercise during chemotherapy for breast cancer. Support Care Cancer. 2020 May;28(5):2115-2126. doi: 10.1007/s00520-019-05019-1. Epub 2019 Aug 8. PMID 31396745
- [Background] Hiraoui M, Al-Haddabi B, Gmada N, Doutrellot PL, Mezlini A, Ahmaidi S. Effects of combined supervised intermittent aerobic, muscle strength and home-based walking training programs on cardiorespiratory responses in women with breast cancer. Bull Cancer. 2019 Jun;106(6):527-537. doi: 10.1016/j.bulcan.2019.03.014. Epub 2019 May 20. PMID 31122656
- [Background] Indelicato DJ, Keole SR, Shahlaee AH, Shi W, Morris CG, Gibbs CP Jr, Scarborough MT, Marcus RB Jr. Long-term clinical and functional outcomes after treatment for localized Ewing's tumor of the lower extremity. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):501-9. doi: 10.1016/j.ijrobp.2007.06.032. Epub 2007 Sep 12. PMID 17855013
- [Background] Mavrogenis AF, Abati CN, Romagnoli C, Ruggieri P. Similar survival but better function for patients after limb salvage versus amputation for distal tibia osteosarcoma. Clin Orthop Relat Res. 2012 Jun;470(6):1735-48. doi: 10.1007/s11999-011-2238-7. Epub 2012 Jan 24. PMID 22270466
- [Background] Morri M, Raffa D, Barbieri M, Ferrari S, Mariani E, Vigna D. Compliance and satisfaction with intensive physiotherapy treatment during chemotherapy in patients with bone tumours and evaluation of related prognostic factors: An observational study. Eur J Cancer Care (Engl). 2018 Nov;27(6):e12916. doi: 10.1111/ecc.12916. Epub 2018 Sep 27. PMID 30260524
- [Background] Carty CP, Bennett MB, Dickinson IC, Steadman P. Assessment of kinematic and kinetic patterns following limb salvage procedures for bone sarcoma. Gait Posture. 2009 Nov;30(4):547-51. doi: 10.1016/j.gaitpost.2009.08.234. Epub 2009 Sep 10. PMID 19747830
- [Background] de Visser E, Deckers JA, Veth RP, Schreuder HW, Mulder TW, Duysens J. Deterioration of balance control after limb-saving surgery. Am J Phys Med Rehabil. 2001 May;80(5):358-65. doi: 10.1097/00002060-200105000-00007. PMID 11327558
- [Background] Rossi L, Boffano M, Comandone A, Ferro A, Grignani G, Linari A, Pellegrino P, Piana R, Ratto N, Davis AM. Validation process of Toronto Exremity Salvage Score in Italian: A quality of life measure for patients with extremity bone and soft tissue tumors. J Surg Oncol. 2020 Mar;121(4):630-637. doi: 10.1002/jso.25849. Epub 2020 Jan 19. PMID 31957034
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Bahcaci U, Demirbuken I. Effects of chemotherapy process on postural balance control in patients with breast cancer. Indian J Cancer. 2019 Jan-Mar;56(1):50-54. doi: 10.4103/ijc.IJC_47_18. PMID 30950445